CLINICAL TRIAL: NCT07250178
Title: Effect of Surgical Approach on Optic Nerve Sheath Diameter as a Surrogate Marker of Intracranial Pressure: A Comparison Between vNOTES and Total Laparoscopic Hysterectomy
Brief Title: ONSD as an ICP Marker in vNOTES and TLH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Acil,MD, Principal Investigator, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/05/2025-627
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer; Abnormal Uterine Bleeding; Myoma;Uterus
Keywords: Laparoscopic Hysterectomy; vNOTES; Optic Nerve Sheath Diameter; Intracranial Pressure
MeSH Terms: conditions — Endometrial Neoplasms; Metrorrhagia; Myofibroma

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, randomized controlled trial with a parallel assignment design. Eligible patients undergoing elective laparoscopic hysterectomy will be randomly allocated in a 1:1 ratio to either the vNOTES group or the TLH group. Randomization will be performed using a computer-generated sequence, and allocation concealment will be maintained with sealed opaque envelopes. Each participant will receive only one surgical intervention.
Masking Description: Due to the nature of the surgical interventions, blinding is not feasible. Both surgeons and outcome assessors are aware of group allocation. Participants may also recognize their assigned intervention based on the operative approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vNOTES Hysterectomy for Assessment of Intraoperative Optic Nerve Sheath Diameter (Experimental): Vajinal natural orifice transluminal endoscopic surgery (vNOTES): In the vNOTES group, the surgery was performed using a transvaginal approach with a self-retaining vaginal port. Following colpotomy, CO₂ insufflation was applied through the vaginal port, ensuring intra-abdominal pressure did not exceed 15 mmHg. The procedure involved occlusion and ligation of the uterine artery under direct endoscopic visualization, followed by sampling through the vaginal route. Pneumoperitoneum was released before closing the vaginal vault. The uterus was then removed through the vaginal route.
  Interventions: Procedure: vNOTES
- Total Laparoscopic Hysterectomy for Assessment of Intraoperative Optic Nerve Sheath Diameter (Active Comparator): Total laparoscopic hysterectomy (TLH): In the TLH group, the surgical procedure was performed under standard laparoscopic conditions using a 10 mm umbilical camera port and two 5 mm accessory trocars. CO₂ insufflation was initiated to maintain intra-abdominal pressure below 15 mmHg. The uterus is dissected using a bipolar vessel sealing device, and the specimen is removed transvaginally. The vaginal cuff and abdominal trocar entries are sutured laparoscopically under direct visualization.
  Interventions: Procedure: TLH

INTERVENTIONS:
Procedure: vNOTES — vNOTES: In the vNOTES group, the surgery was performed using a transvaginal approach with a self-retaining vaginal port. Following colpotomy, CO₂ insufflation was applied through the vaginal port, ensuring intra-abdominal pressure did not exceed 15 mmHg. The procedure involved occlusion and ligation of the uterine artery under direct endoscopic visualization, followed by sampling through the vaginal route. Pneumoperitoneum was released before closing the vaginal vault. The uterus was then removed through the vaginal route.
  Arms: vNOTES Hysterectomy for Assessment of Intraoperative Optic Nerve Sheath Diameter
Procedure: TLH — In the TLH group, the surgical procedure was performed under standard laparoscopic conditions using a 10 mm umbilical camera port and two 5 mm accessory trocars. CO₂ insufflation was initiated to maintain intra-abdominal pressure below 15 mmHg. The uterus is dissected using a bipolar vessel sealing device, and the specimen is removed transvaginally. The vaginal cuff and abdominal trocar entries are sutured laparoscopically under direct visualization.
  Arms: Total Laparoscopic Hysterectomy for Assessment of Intraoperative Optic Nerve Sheath Diameter

SUMMARY:
Patients undergoing conventional total laparoscopic hysterectomy (TLH) are typically placed in the Trendelenburg position with intraabdominal carbon dioxide (CO₂) insufflation. These factors may contribute to intraoperative complications such as lymphedema, impaired pulmonary function, and increased intracranial pressure.

Vaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES), a novel minimally invasive technique, provides retroperitoneal or transperitoneal access through the vaginal route and offers the potential for shorter operative times and lower intraabdominal pressure requirements.

This study aims to evaluate whether the vNOTES technique can reduce intraoperative and postoperative complications compared with TLH. Particular attention will be given to hemodynamic parameters and changes in optic nerve sheath diameter as an indirect indicator of intracranial pressure.

DETAILED DESCRIPTION:
This study is designed as a single-center, prospective, randomized controlled trial conducted at the Gynecologic Oncology Clinic of Health Sciences University Diyarbakır Gazi Yaşargil Training and Research Hospital. Eligible patients will be women between 18 and 75 years of age, classified as ASA I-II, who are scheduled for elective laparoscopic hysterectomy for gynecologic oncology indications. The study protocol will be initiated after approval by the institutional ethics committee, and written informed consent will be obtained from all participants.

Group vNOTES: Following vaginal exposure with a speculum under general anesthesia, entry will be performed through the posterior vaginal fornix. After posterior colpotomy, the vNOTES port system will be inserted. Pneumoperitoneum will be established with CO₂ insufflation at a maximum pressure of 15 mmHg. The operation will be performed using an endoscopic camera and working channels.

Group TLH: Under general anesthesia, pneumoperitoneum will be created via an umbilical trocar (maximum pressure15 mmHg), followed by placement of 2-3 additional trocars in the lower abdomen. A standard total laparoscopic hysterectomy will then be performed.

Demographic and perioperative data will be collected, including age, diagnosis, ASA score, anesthesia and surgery duration, intraoperative blood loss (by suction and sponge count), total intravenous fluids, systolic and diastolic blood pressure, heart rate, oxygen saturation, respiratory rate, end-tidal CO₂, intra-abdominal pressure, and ventilatory parameters (PEEP, peak and plateau airway pressures).

The primary outcome will be changes in optic nerve sheath diameter (ONSD), measured by ultrasonography at predefined time points as a surrogate marker of intracranial pressure:

T0: before induction of anesthesia

T1: at 10 minutes after Trendelenburg positioning and insufflation

T2: at 30 minutes

T3: at 60 minutes

T4: at 90 minutes

T5: 10 minutes after desufflation and return to neutral position

All ONSD measurements will be performed intraoperatively by a trained anesthesiologist using standardized ultrasound techniques. Hemodynamic and ventilatory parameters will be recorded at 10-minute intervals.

Secondary outcomes will include arterial blood gas analysis, postoperative complications (such as nausea, vomiting, delirium, headache, dizziness, and diplopia), and recovery variables (time to ambulation, return of bowel function, oral intake, and hospital stay).

Among the parameters measured, ONSD evaluation via ultrasound is specific to the study and non-invasive, adding no risk or cost to the patient. All other parameters are part of routine intraoperative monitoring. Data collection will be carried out in the operating room by anesthesiologists and trained ICU/gynecologic oncology nurses.

The investigators hypothesize that the vNOTES approach, due to its shorter operative duration, reduced Trendelenburg requirements, and lower intraabdominal insufflation pressures, will result in less pronounced increases in ONSD compared with TLH. This may lead to greater intraoperative stability and reduced postoperative complications, thereby providing valuable evidence for optimizing surgical strategies in gynecologic oncology.

ELIGIBILITY:
Inclusion Criteria:

* voluntary participation,
* elective laparoscopic hysterectomy scheduled by gynecology-oncology specialists,
* ASA physical status I-II

Exclusion Criteria:

* included unwillingness to participate,
* emergency surgery,
* age <18 years,
* prior major pelvic or abdominal surgery,
* ASA ≥III,
* Chronic pulmonary disease, pulmonary hypertension, glaucoma, diabetic retinopathy, intracranial pathology (mass, hydrocephalus, optic neuritis), prior ocular or intracranial surgery, cardiac failure (EF <40%), active infection, or systemic inflammatory diseases other than malignancy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female patients are eligible for inclusion, as the surgical procedures under investigation (vNOTES and total laparoscopic hysterectomy) are applicable solely to women undergoing gynecologic surgery.
Enrollment: 66 (Actual)
Dates: Start 2025-11-27 (Actual); Primary Completion 2026-01-02 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter (ONSD) measured | From baseline (before induction) to 10, 30, 60, and 90 minutes after Trendelenburg and CO₂ insufflation, and 10 minutes after desufflation.
  All measurements were performed using a high-resolution ultrasound device equipped with a 7-13 MHz linear probe. The ultrasound gain and depth settings were standardized for all patients (depth: 4-5 cm; focus: at the level of the optic disc). Patient Position: Measurements were obtained with patients in the supine position. The eyes were kept closed, and sterile ultrasound gel was applied without exerting pressure on the globe. The probe was gently placed on the upper eyelid, and measurements were taken in the transverse plane. The optic nerve sheath diameter was measured 3 mm distal to the optic disc, from outer edge to outer edge (outer-to-outer).

SECONDARY OUTCOMES:
Blood pressure measurement | It will be recorded 10 minutes before induction of anesthesia and every 15 minutes after intubation until the end of the operation.
  Systolic, diastolic and mean arterial pressure measurements will be recorded by invasive arterial monitoring.
Measurement of heart rate | It will be recorded 10 minutes before induction of anesthesia and every 15 minutes after intubation until the end of the operation.
  The number of heart beats per minute obtained by electrocardiographic monitoring
intraabdominal pressure | It will be recorded 10 minutes before induction of anesthesia and every 15 minutes after intubation until the end of the operation.
  The pressure inside the abdominal cavity during CO₂ insufflation.
end-tidal CO₂ (EtCO₂) | It will be recorded 10 minutes before induction of anesthesia and every 15 minutes after intubation until the end of the operation.
  The partial pressure of CO₂ at end-expiration measured by capnography
peak airway pressure | It will be recorded 10 minutes before induction of anesthesia and every 15 minutes after intubation until the end of the operation.
  The highest pressure reached in the airways during inspiration under mechanical ventilation.
Nausea-vomiting | During the 24 hours postoperative period
  Questioning about the presence/absence of nausea and/or vomiting in the postoperative period
dizziness | During the 24 hours postoperative period
  Questioning about the presence/absence of dizzines the postoperative period
diplopia | During the 24 hours postoperative period
  Questioning about the presence/absence of diplopia the postoperative period
Incidence of Postoperative Headache | Within the first 24 hours postoperatively
  The incidence of postoperative headache will be recorded within the first 24 hours after surgery. Headache will be assessed by direct patient questioning and documented as present or absent.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Acil, M.D., Principal Investigator — Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Locations (1):
- Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital, Diyarbakır, Outside of the US, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including baseline demographic variables and primary/secondary outcome measures, will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: study completion + 6 months
Access Criteria: Researchers may request access to the de-identified IPD by contacting the principal investigator at:[acilfatma@gmail.com].
  Requests will be evaluated by the investigators, and data will be shared after approval and completion of a data-sharing agreement."

REFERENCES:
- [Background] Guloglu H, Cetinkaya D, Oge T, Bilir A. Evaluation of the effect of trendelenburg position duration on intracranial pressure in laparoscopic hysterectomies using ultrasonographic optic nerve sheath diameter measurements. BMC Anesthesiol. 2024 Jul 15;24(1):238. doi: 10.1186/s12871-024-02624-4. PMID 39010013